CLINICAL TRIAL: NCT01512706
Title: A Phase II Clinical Trial for Inactivated Enterovirus Type 71 Vaccine (Human Diploid Cell, KMB-17 Cell) in Chinese Infants
Brief Title: A Phase II, Safety and Efficacy Study of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Guangxi Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EV71-KMB17-II-IMB-CAMS
Record Dates: First submitted 2012-01-15; First posted 2012-01-19 (Estimated); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: The Study Focused on the Safety of Inactivated EV71 Vaccine (Human Diploid Cell) Against Hand, Foot and Mouth Disease in Chinese Children and Infants
Keywords: Human Enterovirus 71 (EV71); Hand, Foot and Mouth Disease; Inactivated Vaccine; Human Diploid cell; Safety; Immunogenicity; Adverse reactions associated with vaccine
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- 160Eu/0.5ml in infants (6-11 months old) (Experimental): inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 60 infants aged 6-11 months old on day 0, 28
  Interventions: Biological: 160Eu/0.5ml in infants (6-11 months old)
- 320Eu/0.5ml in infants (6-11 months old) (Experimental): inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 60 infants aged 6-11 months old on day 0, 28
  Interventions: Biological: 320Eu/0.5ml in infants (6-11 months old)
- 640Eu/0.5ml in infants (6-11 months old) (Experimental): inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 40 infants aged 6-11 months old on day 0, 28
  Interventions: Biological: 640Eu/0.5ml in infants (6-11 months old)
- 1280Eu/0.5ml in infants (6-11 months old) (Experimental): inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 40 infants aged 6-11 months old on day 0, 28
  Interventions: Biological: 1280Eu/0.5ml (without adjuvant) in infants (6-11 months old)
- 0Eu/0.5ml in infants (6-11 months old) (Placebo Comparator): 0Eu/0.5ml placebo in 80 infants aged 6-11 months old on day 0, 28
  Interventions: Biological: 0Eu/0.5ml in infants (6-11 months old)
- 160Eu/0.5ml in infants (12-23 months old) (Experimental): inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 30 infants aged 12-23 months old on day 0, 28
  Interventions: Biological: 160Eu/0.5ml in infants (12-23 months old)
- 320Eu/0.5ml in infants (12-23 months old) (Experimental): inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 30 infants aged 12-23 months old on day 0, 28
  Interventions: Biological: 320Eu/0.5ml in infants (12-23 months old)
- 640Eu/0.5ml in infants (12-23 months old) (Experimental): inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 40 infants aged 12-23 months old on day 0, 28
  Interventions: Biological: 640Eu/0.5ml in infants (12-23 months old)
- 1280Eu/0.5ml in infants (12-23 months old) (Experimental): inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 40 infants aged 12-23 months old on day 0, 28
  Interventions: Biological: 1280Eu/0.5ml (without adjuvant) in infants (12-23 months old)
- 0Eu/0.5ml in infants (12-23 months old) (Placebo Comparator): 0Eu/0.5ml placebo in 50 infants aged 12-23 months old on day 0, 28
  Interventions: Biological: 0Eu/0.5ml in infants (12-23 months old)
- 160Eu/0.5ml in children (24 months-5 years old) (Experimental): inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 30 children aged 24 months-5 years months old on day 0, 28
  Interventions: Biological: 160Eu/0.5ml in children (24 months-5 years old)
- 320Eu/0.5ml in children (24 months-5 years old) (Experimental): inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 30 children aged 24 months-5 years months old on day 0, 28
  Interventions: Biological: 320Eu/0.5ml in children (24 months-5 years old)
- 640Eu/0.5ml in children (24 months-5 years old) (Experimental): inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 40 children aged 24 months-5 years months old on day 0, 28
  Interventions: Biological: 640Eu/0.5ml in children (24 months-5 years old)
- 1280Eu/0.5ml in children (24 months-5 years old) (Experimental): inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 40 children aged 24 months-5 years months old on day 0, 28
  Interventions: Biological: 1280Eu/0.5ml (without adjuvant) in children (24 months-5 years old)
- 0Eu/0.5ml in children (24 months-5 years old) (Placebo Comparator): 0Eu/0.5ml placebo in 50 children aged 24 months-5 years old on day 0, 28
  Interventions: Biological: 0Eu/0.5ml in children (24 months-5 years old)

INTERVENTIONS:
Biological: 160Eu/0.5ml in infants (6-11 months old) — inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 60 infants aged 6-11 months old on day 0, 28
  Arms: 160Eu/0.5ml in infants (6-11 months old)
Biological: 320Eu/0.5ml in infants (6-11 months old) — inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 60 infants aged 6-11 months old on day 0, 28
  Arms: 320Eu/0.5ml in infants (6-11 months old)
Biological: 640Eu/0.5ml in infants (6-11 months old) — inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 40 infants aged 6-11 months old on day 0, 28
  Arms: 640Eu/0.5ml in infants (6-11 months old)
Biological: 1280Eu/0.5ml (without adjuvant) in infants (6-11 months old) — inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 40 infants aged 6-11 months old on day 0, 28
  Arms: 1280Eu/0.5ml in infants (6-11 months old)
Biological: 0Eu/0.5ml in infants (6-11 months old) — 0Eu/0.5ml placebo in 80 infants aged 6-11 months old on day 0, 28
  Arms: 0Eu/0.5ml in infants (6-11 months old)
Biological: 160Eu/0.5ml in infants (12-23 months old) — inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 30 infants aged 12-23 months old on day 0, 28
  Arms: 160Eu/0.5ml in infants (12-23 months old)
Biological: 320Eu/0.5ml in infants (12-23 months old) — inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 30 infants aged 12-23 months old on day 0, 28
  Arms: 320Eu/0.5ml in infants (12-23 months old)
Biological: 640Eu/0.5ml in infants (12-23 months old) — inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 40 infants aged 12-23 months old on day 0, 28
  Arms: 640Eu/0.5ml in infants (12-23 months old)
Biological: 1280Eu/0.5ml (without adjuvant) in infants (12-23 months old) — inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml (without adjuvant) in 40 infants aged 12-23 months old on day 0, 28
  Arms: 1280Eu/0.5ml in infants (12-23 months old)
Biological: 0Eu/0.5ml in infants (12-23 months old) — 0Eu/0.5ml placebo in 50 infants aged 12-23 months old on day 0, 28
  Arms: 0Eu/0.5ml in infants (12-23 months old)
Biological: 160Eu/0.5ml in children (24 months-5 years old) — inactivated EV71 vaccine (KMB-17) of 160Eu/0.5ml in 30 children aged 24 months-5 years months old on day 0, 28
  Arms: 160Eu/0.5ml in children (24 months-5 years old)
Biological: 320Eu/0.5ml in children (24 months-5 years old) — inactivated EV71 vaccine (KMB-17) of 320Eu/0.5ml in 30 children aged 24 months-5 years months old on day 0, 28
  Arms: 320Eu/0.5ml in children (24 months-5 years old)
Biological: 640Eu/0.5ml in children (24 months-5 years old) — inactivated EV71 vaccine (KMB-17) of 640Eu/0.5ml in 40 children aged 24 months-5 years months old on day 0, 28
  Arms: 640Eu/0.5ml in children (24 months-5 years old)
Biological: 1280Eu/0.5ml (without adjuvant) in children (24 months-5 years old) — inactivated EV71 vaccine (KMB-17) of 1280Eu/0.5ml in 40 children aged 24 months-5 years months old on day 0, 28
  Arms: 1280Eu/0.5ml in children (24 months-5 years old)
Biological: 0Eu/0.5ml in children (24 months-5 years old) — 0Eu/0.5ml placebo in 50 children aged 24 months-5 years old on day 0, 28
  Arms: 0Eu/0.5ml in children (24 months-5 years old)

SUMMARY:
Enterovirus 71 (EV71), a major pathogen that is responsible for causing hand-foot-and-mouth disease (HFMD) worldwide, is a member of the Human Enterovirus species A, family Picornaviridae.

Since the late 1990s, a series of large HFMD epidemics caused by EV71 have been reported in the Asia-Pacific region. Notably, there is evidence that the most severe cases from these epidemic outbreaks are associated with neurological disorders with CNS involvement caused by EV71 infection. Because of these EV71 infection-related public health issues, the research and development of EV71 vaccine candidates have been heavily promoted.

Recently, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, including inactivated vaccine, attenuated vaccine, subunit vaccine, DNA vaccine, epitope peptide vaccine, virus-like particles (VLPs).

Basing on the previous studies of elicited protection in mice and rhesus monkeys, a formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been licensed by SFDA in China, Dec. 2010. The phase I clinical trial was completed, during four months, in Guangxi Province, China. The phase II clinical trial has been carried out, from July 2011. The purpose of phase II is to evaluate the safety and efficacy of the formalin-inactivated EV71 vaccine in Chinese infants (from 6 to 36 months old).

DETAILED DESCRIPTION:
Hand-foot-and-mouth disease (HFMD) is a significant cause of death, usually characterized by vesicular lesions on the skin and oral mucosa and high morbidity rates in children. Additionally, occasional fatal cases have been reported involving brainstem encephalitis and myelitis associated with cardiopulmonary collapse. Pulmonary edema/hemorrhage and respiratory failure are the major causes of death among children less than five years old.

Enterovirus 71 (EV71), a major pathogen that is responsible for causing HFMD worldwide, is a member of the Human Enterovirus species A, family Picornaviridae. Since the late 1990s, a series of large HFMD epidemics caused by EV71 have been reported in the Asia-Pacific region. Notably, there is evidence that the most severe cases from these epidemic outbreaks are associated with neurological disorders with CNS involvement caused by EV71 infection. Because of these EV71 infection-related public health issues, the research and development of EV71 vaccine candidates have been heavily promoted.

Recently, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, including heat-inactivated or formalin-inactivated vaccine, live-attenuated vaccine, recombinant viral protein 1 (VP1) vaccine, VP1 DNA vaccine, VP1 epitope peptide vaccine, EV71 virus-like particles (VLPs) and bacterial or viral vector expressing VP1. Overall, the inactivated whole-virus vaccines seem to be more immunogenic than recombinant VP1 and DNA vaccines.

Basing on the previous studies of elicited protection in mice and rhesus monkeys (Ying Zhang, et al. Pathogenesis study of Enterovirus 71 Infection in Rhesus Monkeys. Lab Invest, 2011, doi:10.1038/labinest.2011.82; Longding Liu, et al. Neonatal Rhesus Monkey is a Potential Animal Model for Studying Pathogenesis of EV71 Infection. Virology, 2011, 412:91-100; Chenghong Dong, et al. Immunoprotection Elicited by an Enterovirus Type 71 Experimental Inactivated Vaccine in Mice and Rhesus Monkeys. Vaccine, 2011, doi: 10.1016/j.vaccine.2011.06.044.), a formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been licensed by SFDA in China, Dec. 2010. The phase I clinical trial was completed, during four months, in Guangxi Province, China.

The results showed that the formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) was safety in Chinese adults (from 18 to 49 years old), children (from 3 to 11 years old) and infants (from 6 to 35 months old). This vaccine could induce specific cellular and humoral immune responses.

The phase II clinical trial has been carried out, from July 2011. The purpose of phase II is to evaluate the safety and efficacy of the formalin-inactivated EV71 vaccine in Chinese infants (from 6 to 36 months old).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (6-35 months infants) as established by medical history and clinical examination
* Full-term (37-42 weeks), weight ≥ 2500 g when it was born
* The subjects' legal guardian must be aware of this vaccines
* The subjects' legal guardian voluntarily participate in the study and signed Informed Consent Form
* Subjects with temperature ≤ 37.0℃
* The subjects' legal guardian with the ability and objective to comply with the requirements of the protocol
* Persist for a 2-month visit and receive blood tests according to program requirements

Exclusion Criteria:

* Subject who has a clinical diagnosis history of Hand, Foot and Mouth Disease (HFMD)

  * 37 weeks gestation
* weight ≤ 2500 g when it was born
* Allergy or serious side-effects to a vaccine or any ingredient of vaccine
* Epilepsy, seizures, convulsions, neurological illness
* Congenital or hereditary immunodeficiency
* Autoimmune disease
* Severe malnutrition or dysgenopathy
* Asthma, thyroidectomy, angioneurotic edema, diabetes or cancer
* Asplenia, functional asplenia, and any circumstances leading to the asplenia or splenectomy
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder
* Acute illness or acute exacerbation of chronic disease in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of live-attenuated vaccine in last 28 days or 1 months
* Any prior administration of subunit or inactivated vaccines in last 14 days Under the anti-TB prevention or therapy
* Fever before vaccination, axillary temperature ﹥37.0℃
* The laboratory test abnormalities before vaccination, including blood tests (hemoglobin, total white blood cells, WBC, platelets), blood biochemistry tests (ALT, total bilirubin, direct bilirubin, Cr, BUN) and urine tests (urine protein, urine sugar, blood cells), etc.
* Hypertension or hypotension. Systolic blood pressure ﹥140mmHg and/or diastolic blood pressure ﹥90mmHg; systolic blood pressure ﹤90mmHg and/or diastolic blood pressure ﹤60mmHg
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 660 (Actual)
Dates: Start 2011-07; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants (from 6 to 11 months old) | within the first 28 days after the first vaccination
  Adverse reactions associated with vaccine were observed in Chinese Infants (from 6 to 11 months old) after the first vaccination.
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants (from 12 to 23 months old) | within the first 28 days after the first vaccination
  Adverse reactions associated with vaccine were observed in Chinese Infants (from 12 to 23 months old) after the first vaccination
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese children (from 24 months to 5 years old) | within the first 28 days after the first vaccination
  Adverse reactions associated with vaccine were observed in Chinese children (from 24 months to 5 years old) after the first vaccination
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants (from 6 to 11 months old) | within the first 56 days after the second vaccination
  Adverse reactions associated with vaccine were observed in Chinese Infants (from 6 to 11 months old) after the second vaccination
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese Infants (from 12 to 23 months old) | within the first 56 days after the second vaccination
  Adverse reactions associated with vaccine were observed in Chinese Infants (from 12 to 23 months old) after the second vaccination
Evaluate the safety of Inactivated EV 71 Vaccine (Human Diploid Cell, KMB-17) in Chinese children (from 24 months to 5 years old) | within the first 56 days after the second vaccination
  Adverse reactions associated with vaccine were observed in Chinese children (from 24 months to 5 years old) after the second vaccination

SECONDARY OUTCOMES:
Evaluate the seroconversion rate of anti-EV71 antibodies in serum of children and infant, after first vaccination | at the 28 day after the first vaccination
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of children and infant, at the 28 day after the first vaccination
Evaluate the seroconversion rate of anti-EV71 antibodies in serum of children and infant, after second vaccination | at the 28 or 56 days after the second vaccination
  The seroconversion rate of anti-EV71 antibodies was evaluated in serum of children and infant, at the 28 or 56 days after the second vaccination
Evaluate the seroconversion rate of antinuclear antibodies in serum of children and infant, after first vaccination | at the 28 day after the first vaccination
  The seroconversion rate of antinuclear antibodies was evaluated in serum of children and infant, at the 28 day after the first vaccination
Evaluate the seroconversion rate of antinuclear antibodies in serum of children and infant, after second vaccination | at the 28 or 56 days after the second vaccination
  The seroconversion rate of antinuclear antibodies was evaluated in serum of children and infant, the 28 or 56 days after the second vaccination
Evaluate the abnormity change of live and kidney function indexes in serum of children and infant, after first vaccination | at the 28 days after the first vaccination
  The abnormity change of live and kidney function indexes were evaluated in serum of children and infant, at the 28 days after the first vaccination
Evaluate the abnormity change of live and kidney function indexes in serum of children and infant, after second vaccination | at the 28 or 56 days after the second vaccination
  The abnormity change of live and kidney function indexes were evaluated in serum of children and infant, the 28 or 56 days after the second vaccination
Evaluate the abnormity change of body temperature of children and infant, after first vaccination | within the first 28 days after the first vaccination
  The abnormity change of body temperature of children and infant were evaluated, at the 28 days after the first vaccination
Evaluate the abnormity change of body temperature of children and infant, after second vaccination | within the first 56 days after the second vaccination
  The abnormity change of body temperature of children and infant were evaluated, within the first 56 days after the second vaccination
Evaluate the vaccine-induced cellular immune responses in children and infant after first vaccination | at the 28 day after the first vaccination
  The vaccine-induced cellular immune responses were evaluated in serum of children and infant, at the 28 day after the first vaccination
Evaluate the vaccine-induced cellular immune responses in children and infant after second vaccination | at the 28 or 56 days after the second vaccination
  The vaccine-induced cellular immune responses were evaluated in serum of children and infant, at the 28 or 56 days after the second vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Zhaojun Mo, Master, Principal Investigator — Guangxi Provincial Center for Diseases Control and Prevention
Locations (1):
- Guangxi Provincial Center for Diseases Control and Prevention, Nanning, Guangxi, China

REFERENCES:
- [Derived] Zhang Y, Wang L, Liao Y, Liu L, Ma K, Yang E, Wang J, Che Y, Jiang L, Pu J, Guo L, Feng M, Liang Y, Cui W, Yang H, Li Q. Similar protective immunity induced by an inactivated enterovirus 71 (EV71) vaccine in neonatal rhesus macaques and children. Vaccine. 2015 Nov 17;33(46):6290-7. doi: 10.1016/j.vaccine.2015.09.047. Epub 2015 Sep 28. PMID 26419198
- [Derived] Liu L, Zhang Y, Wang J, Zhao H, Jiang L, Che Y, Shi H, Li R, Mo Z, Huang T, Liang Z, Mao Q, Wang L, Dong C, Liao Y, Guo L, Yang E, Pu J, Yue L, Zhou Z, Li Q. Study of the integrated immune response induced by an inactivated EV71 vaccine. PLoS One. 2013;8(1):e54451. doi: 10.1371/journal.pone.0054451. Epub 2013 Jan 23. PMID 23372725